CLINICAL TRIAL: NCT01896518
Title: Novel Methods to Reduce Children's Secondhand Smoke Exposure II
Acronym: EZII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0642; 1R21CA164521-01A1 (NIH)
Record Dates: First submitted 2013-06-20; First posted 2013-07-11 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Secondhand Smoke
Keywords: second hand smoke exposure; children
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Counseling (No Intervention)
- Nicotine lozenge (Experimental): Participants will receive nicotine lozenge to use as needed for 12 weeks.
  Interventions: Drug: Nicotine polacrilex
- Tobacco lozenge (Experimental): Participants will receive tobacco lozenge to use as needed for 12 weeks.
  Interventions: Drug: Tobacco lozenge

INTERVENTIONS:
Drug: Nicotine polacrilex
  Arms: Nicotine lozenge
Drug: Tobacco lozenge
  Arms: Tobacco lozenge

SUMMARY:
The overall aim of the current study is to determine if the use of nicotine containing products by caregivers who smoke and who are not interested in quitting, is effective in reducing children's secondhand smoke exposure.

ELIGIBILITY:
Inclusion Criteria:

In order to be included in the study, participants must:

1. be the primary caregiver(defined as a person who spends the most time with the child and spends a minimum of 4 hours per day in the presence of the child) of a child between the ages of 3-11 (if caregiver has more > 1 child between 3-11 years, we will include the youngest),
2. smoke at least 10 cigarettes per day for the past year,
3. indicate that they smoke around their child or in the car or home at least one time per week],
4. have no intention of quitting smoking in the next 12-weeks,
5. aged 18-65 years,
6. be fluent in English,
7. have no recent history of cardiovascular distress that may contraindicate medicinal nicotine lozenge use (heart attack in the past year, arrhythmia, uncontrolled hypertension),
8. not currently pregnant, planning to become pregnant, or breastfeeding,
9. do not use non-cigarette tobacco (cigars, chewing tobacco)
10. have no prior use of any potential reduced exposure product,
11. have no major psychiatric impairment, including psychosis, suicidality, and/or any current alcohol/drug abuse or dependence

Exclusion Criteria:

Does not meet all of the requirements of inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Child Salivary Cotinine | 3, 6, and 12 weeks
  Child salivary cotinine will be measured to assess the level of secondhand smoke exposure. We will measure the change throughout the study.

SECONDARY OUTCOMES:
Change in Parent and Child Lung Function | 3, 6, 12 weeks
  We will collect both parent and child spirometry data and compare changes.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Wagener, Ph.D., Principal Investigator — OTRC, OU Children's Hospital Dept. of Pediatrics, OU Cancer Center
Locations (1):
- The Children's Hospital at OU Medical Center, Oklahoma City, Oklahoma, United States